CLINICAL TRIAL: NCT03235544
Title: A Phase 2, Open-Label, 2-Cohort, Multicenter Study of INCB050465, a PI3Kδ Inhibitor, in Relapsed or Refractory Mantle Cell Lymphoma Previously Treated With or Without a BTK Inhibitor (CITADEL-205)
Brief Title: A Study of INCB050465 in Relapsed or Refractory Mantle Cell Lymphoma Previously Treated With or Without a Bruton's Tyrosine Kinase (BTK) Inhibitor
Acronym: (CITADEL-205)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-205 (CITADEL-205); Parsaclisib (Other: Incyte Corporation); 2017-003148-19 (EudraCT Number)
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma
Keywords: Mantle cell lymphoma; non-Hodgkin lymphoma; Bruton's tyrosine kinase (BTK); phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Treatment A (Exposed to Ibrutinib) (Experimental): Participants received parsaclisib 20 mg tablets, orally, once daily (QD) for 8 weeks followed by 20 mg once weekly (QW) for up to 52 weeks.
  Participants who were exposed to ibrutinib before enrollment were included in this group.
  Interventions: Drug: Parsaclisib
- Cohort 1: Treatment B (Exposed to Ibrutinib) (Experimental): Participants received parsaclisib 20 mg tablets, orally, QD for 8 weeks followed by 2.5 mg QD for up to 116 weeks.
  Participants who were exposed to ibrutinib before enrollment were included in this group.
  Interventions: Drug: Parsaclisib
- Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) (Experimental): Participants received parsaclisib 20 mg tablets, orally, QD for 8 weeks followed by 20 mg QW for up to approximately 145 weeks.
  Participants who had not received a BTK inhibitor previously were included in this group.
  Interventions: Drug: Parsaclisib
- Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve) (Experimental): Participants received parsaclisib 20 mg tablets, orally, QD for 8 weeks followed by 2.5 mg QD for up to approximately 136 weeks.
  Participants who had not received a BTK inhibitor previously were included in this group.
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib tablets administered orally with water and without regard to food.
  Other Names: INCB050465

SUMMARY:
This is a Phase 2, open-label, 2-cohort study designed to evaluate the efficacy and safety of 2 parsaclisib treatment regimens in participants with relapsed or refractory mantle cell lymphoma (MCL) previously treated either with or without a Bruton's tyrosine kinase (BTK) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 years or older.
* Documented failure to achieve at least partial response (PR) with, or documented disease progression after, the most recent treatment regimen.
* Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.

Exclusion Criteria:

* History of central nervous system lymphoma (either primary or metastatic).
* Prior treatment with idelalisib, other selective phosphatidylinositol 3-kinase delta (PI3Kδ) inhibitors, or a pan PI3K inhibitor.
* Allogeneic stem cell transplant within the last 6 months, or autologous stem cell transplant within the last 3 months before the date of first dose of study treatment.
* Active graft-versus-host disease.
* Liver disease: Participants positive for hepatitis B surface antigen or hepatitis B core antibody will be eligible if they are negative for hepatitis B virus-deoxyribonucleic acid (HBV-DNA). Participants positive for anti-hepatitis C virus (HCV) antibody will be eligible if they are negative for HCV-ribonucleic acid (RNA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, Study Director — Incyte Corporation
Locations (103):
- United States (21):
  - University of Alabama At Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Rocky Mountain Cancer Center-Aurora, Aurora, Colorado
  - Asclepes Research Centers, Brooksville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Bond & Steele Clinic, P.A., Winter Haven, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Hattiesburg Clinic Hematology, Hattiesburg, Mississippi
  - Clinical Research Alliance, Inc., New Hyde Park, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Kaiser Permanente - Northwest, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Texas Oncology, Austin, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Yakima Valley Memorial Hospital/North Star, Yakima, Washington
- Belgium (4):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Institut Jules Bordet, Brussels
  - Hopital de Jolimont, La Louvière
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- Czechia (4):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Kralovske Vinohadry, Interni Hematologicka Klinika, Prague
  - Charles University General Hospital, Prague
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus Universitets Hospital, Aarhus
  - Odense Universitetshospital (Ouh) (Odense University Hospital), Odense C
  - Zealand University Hospital, Roskilde
- France (16):
  - Avicenne Hospital, Bobigny
  - Chu de Clermont - Ferrand- Hospital Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - University Hospital Grenoble, Grenoble
  - Centre Hospitalier Departemental - La-Roche-Sur-Yon - Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint-Louis, Paris
  - H�Pital Universitaire Piti�-Salp�Tri�Re, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Henri Becquerel, Rouen
  - Chru Hopitaux de Tours, Hospital Bretonneau, Tours
  - Institute Gustave Roussy (Igr), Villejuif
- Germany (8):
  - Praxis Brudler, Heinrich, Bangerter, Augsburg
  - Universitaetsklinikum Essen, Essen
  - Universit�Tsklinikum Essen, Essen
  - Justus-Liebig University, Giessen
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Kliniken Maria Hilf, Mönchengladbach
  - Rotkreuzklinikum Munich, München
  - Universit�Tsklinikum Ulm, Ulm
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan, MI
  - Centro Ricerche Cliniche, Bologna
  - Azienda Policlinico Vittorio Emanuele, Catania
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Niguarda Ca Granda, Milan
  - A.O.U. Di Modena - Policlinico, Modena
  - A.O.U. Federico Ii, Napoli
  - Aou Maggiore Della Carita, Novara
  - Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Sapienza University, Rome
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria Alle Scotte, Siena
  - Azienda Ospedaliero Universitaria Citta Della Salute E Della Scienza, Torino
- Poland (6):
  - Beskidzkie Centrum Onkologii Im.Jana Pawla Ii, Bielsko-Biala
  - Szpital Specjalistyczny W Brzozowie, Podkarpacki Osrodek Onkologiczny Im.Ks.B.Markiewicza, Brzozów
  - University Clinical Center, Gdansk
  - Pratia McM Krakow, Krakow
  - Nu-Med Centrum Diagnostykii I Terapii Onkologicznej, Tomaszów Mazowiecki
  - Centrum Onkologii-Instytut Im. Marii Sklodowskiej-Curie, Warsaw
- Spain (18):
  - Hospital Del Mar, Barcelona
  - Hospital General Universitari Vall D Hebron, Barcelona
  - Hospital Universitari Mutua Terrassa, Barcelona
  - Institut Catala D Oncologia, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Md Anderson Cancer Centre Madrid, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario Y Politecnic La Fe, Valencia
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - Western General Hospital, Edinburgh
  - University College London Hospitals (Uclh), London
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available to interested researchers after the end of study, a thorough analysis, and the publication of the data in the clinical study report (CSR). As required, results of the data will be posted to ClinicalTrials.gov. Upon request, individual investigators may obtain IPD from the sponsor. The format for data delivery will be determined between sponsor and investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 76 investigative sites in France, Spain, the United States, Italy, Poland, Czech Republic, Great Britain, Denmark, Belgium, Germany, and Israel.
Pre-assignment Details: A total of 161 participants with relapsed or refractory mantle cell lymphoma who received 1-3 prior systemic therapies were enrolled into 2 Cohorts and treated. An additional participant was enrolled but not treated. Because this participant was not treated, he/she was not assigned to any treatment/cohort and was not included in the "Full Analysis Set" or "Safety Population" for analysis. Cohort 1 had previously received ibrutinib and Cohort 2 were Bruton's tyrosine kinase (BTK) inhibitor naive.
Groups:
- Cohort 1: Treatment A (Exposed to Ibrutinib): Participants received parsaclisib 20 milligrams (mg), orally, once daily (QD) for 8 weeks followed by 20 mg once weekly (QW) for up to 52 weeks. Participants who were exposed to ibrutinib before enrollment were included in this group.
- Cohort 1: Treatment B (Exposed to Ibrutinib): Participants received parsaclisib 20 mg, orally, QD for 8 weeks followed by 2.5 mg QD for up to 116 weeks. Participants who were exposed to ibrutinib before enrollment were included in this group.
- Cohort 2: Treatment A (BTK Inhibitor Naïve): Participants received parsaclisib 20 mg, orally, QD for 8 weeks followed by 20 mg QW for up to approximately 145 weeks. Participants who were not exposed to BTK inhibitor before enrollment were included in this group.
- Cohort 2: Treatment B (BTK Inhibitor Naïve): Participants received parsaclisib 20 mg, orally, QD for 8 weeks followed by 2.5 mg QD for up to approximately 136 weeks. Participants who were not exposed to BTK inhibitor before enrollment were included in this group.
Period: Overall Study
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Started | 12 | 41 | 31 | 77
Completed | 1 | 5 | 8 | 29
Not Completed | 11 | 36 | 23 | 48
Not completed — Death | 11 | 31 | 19 | 34
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 5
Not completed — Disease Progression | 0 | 1 | 0 | 2
Not completed — Participant Transitioned to Rollover Protocol | 0 | 0 | 2 | 5
Not completed — Discomfort, Pain, and Radiographic Advancement | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of parsaclisib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve) | Total
Number analyzed (Participants) | 12 | 41 | 31 | 77 | 161
Age, Continuous [Mean (Full Range); unit: years] | 70.2 [53 to 82] | 69.8 [48 to 89] | 72.2 [43 to 89] | 71.5 [51 to 90] | 70.9 [43 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 5 | 17 | 34
  Male | 11 | 30 | 26 | 60 | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 4 | 5 | 14
  Not Hispanic or Latino | 6 | 28 | 21 | 57 | 112
  Not Reported | 1 | 5 | 6 | 8 | 20
  Unknown | 2 | 4 | 0 | 1 | 7
  Captured as "Other" in Database | 0 | 0 | 0 | 2 | 2
  Missing | 0 | 2 | 0 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 37 | 24 | 64 | 136
  Black or African American | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 0 | 1 | 1
  American-Indian/Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0
  Captured as "Other" in Database | 1 | 1 | 5 | 3 | 10
  Missing | 0 | 3 | 2 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR=percentage of participants with complete response(CR) or partial response(PR) per revised response criteria for lymphomas,determined by independent review committee(IRC).Criteria for CR:1.Target nodes/nodal masses of lymph nodes,extralymphatic sites regressed to≤1.5cm in longest dimension transverse diameter of lesion(LDi);2.Absence of non-measured lesion;3.Organ enlargement regressed to normal;4.No new lesions;5.Normal bone marrow morphology;if indeterminate,immunohistochemistry negative.Criteria for PR:1.Lymph nodes,extralymphatic sites- ≥50%decrease in sum of product of perpendicular diameters for multiple lesions(SPD)of up to 6 target measurable nodes,extranodal sites;if lesion is too small to measure on computed tomography(CT),assign5mm×5mm as default;if no longer visible,0×0mm.Node>5mm×5mm but smaller than normal,use actual measurement.2.Absent/regressed non-measured lesions,no increase.3.Organ enlargement-Spleen regressed by>50%in length beyond normal.4.No new lesions.
Time Frame: Up to 1016 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Number analyzed (Participants) | 12 | 41 | 31 | 77
percentage of participants | 8.3 [0.2 to 38.5] | 39.0 [24.2 to 55.5] | 64.5 [45.4 to 80.8] | 71.4 [60.0 to 81.2]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR=time from first documented evidence of CR or PR until disease progression or death from any cause among participants who achieve an objective response as determined by IRC. Criteria for CR: 1.Target nodes/nodal masses of lymph nodes and extralymphatic sites must regress to ≤ 1.5 cm in LDi; 2. Absence of non-measured lesion; 3.Organ enlargement regressed to normal; 4.No new lesions; 5.Bone marrow must be normal by morphology; if indeterminate, immunohistochemistry negative. The criteria for PR included: 1.Lymph nodes and extralymphatic sites- a. ≥50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; b. when a lesion is too small to measure on CT, assign 5 mm×5 mm as the default; c.when no longer visible, 0×0 mm. For a node >5 mm×5 mm but smaller than normal, use actual measurement. 2.Non-measured lesions- Absent/regressed, but no increase. 3. Organ enlargement-Spleen must have regressed by >50% in length beyond normal. 4.No new lesions.
Time Frame: Up to 1016 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib. Only participants with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Number analyzed (Participants) | 1 | 16 | 20 | 55
months | NA [NA to NA] — The median and the lower and upper limits of the 95% confidence interval (CI) were not estimable due to the low number of participants with events of response. | 3.20 [1.87 to 7.95] | 17.45 [3.81 to NA] — The upper limit of the 95% CI was not estimable due to the low number of participants with events of response. | 13.01 [9.03 to 16.59]

3. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of participants with a CR as defined by response criteria for lymphomas, as determined by an IRC. The criteria for CR included: 1.Target nodes/nodal masses of lymph nodes and extralymphatic sites must regress to ≤ 1.5 cm in LDi; 2. Absence of non-measured lesion; 3.Organ enlargement regressed to normal; 4.No new lesions; 5.Bone marrow must be normal by morphology; if indeterminate, immunohistochemistry negative.
Time Frame: Up to 1016 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Number analyzed (Participants) | 12 | 41 | 31 | 77
percentage of participants | 0.0 [0.0 to 26.5] | 2.4 [0.1 to 12.9] | 22.6 [9.6 to 41.1] | 15.6 [8.3 to 25.6]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose of study treatment until the earliest date of disease progression as determined by radiographic disease assessment provided by an IRC, or death from any cause.
Time Frame: Up to 1016 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Number analyzed (Participants) | 12 | 41 | 31 | 77
months | 3.94 [1.35 to NA] — The upper limit of the 95% CI was not estimable due to the low number of participants with events. | 3.68 [1.87 to 5.49] | 8.11 [5.29 to 21.62] | 13.83 [10.02 to 16.89]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose of study treatment until death from any cause.
Time Frame: Up to 2017 days
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Number analyzed (Participants) | 12 | 41 | 31 | 77
months | 10.91 [1.35 to 17.64] | 11.01 [7.23 to 17.12] | 33.48 [21.62 to 54.67] | 45.86 [34.20 to NA] — The upper limit of the confidence interval was not estimable because too few participants died.

6. Secondary Outcome: Best Percent Change From Baseline in Target Lesion Size
Description: Target lesion size is measured by the sum of the product of diameters of all target lesion sizes and is determined by the IRC. The best percent change from Baseline is defined as the largest decrease, or smallest increase if no decrease available, from Baseline in target lesion sizes on/before new (next-line) anti-lymphoma therapy during the study. Baseline is the last nonmissing measurement obtained before the first administration of study drug. A negative percent change from Baseline indicates improvement.
Time Frame: Up to 1016 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib. The overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: percent change in lesion size
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Number analyzed (Participants) | 6 | 32 | 25 | 68
percent change in lesion size | -19.82 (35.926) | -9.51 (133.438) | -64.65 (53.360) | -67.54 (32.918)

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug regardless of starting new anti-lymphoma therapy. A SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect or is considered to be an important medical event that may not result in death, be immediately life-threatening, or require hospitalization but may be considered serious when, based on appropriate medical judgment, the event may jeopardize the participant or may require medical or surgical intervention.
Time Frame: From first dose of study drug up to 2045 days
Population: Safety Population: all enrolled participants who received at least 1 dose of parsaclisib
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve)
Number analyzed (Participants) | 12 | 41 | 31 | 77
percentage of participants
  TEAEs | 83.3 | 90.2 | 93.5 | 92.2
  SAEs | 41.7 | 48.8 | 38.7 | 58.4

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 2045 days
Description: Adverse events have been reported for members of the Safety Population, comprised of all enrolled participants who received at least 1 dose of parsaclisib.
Groups:
- Total: Total
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (BTK Inhibitor Naïve) | Cohort 2: Treatment B (BTK Inhibitor Naïve) | Total
All-Cause Mortality (participants affected / at risk) | 11/12 | 31/41 | 19/31 | 34/77 | 95/161
Serious Adverse Events (participants affected / at risk) | 5/12 | 20/41 | 12/31 | 45/77 | 82/161
Other Adverse Events (participants affected / at risk) | 9/12 | 28/41 | 27/31 | 66/77 | 130/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Treatment A (Exposed to Ibrutinib) (N=12) | Cohort 1: Treatment B (Exposed to Ibrutinib) (N=41) | Cohort 2: Treatment A (BTK Inhibitor Naïve) (N=31) | Cohort 2: Treatment B (BTK Inhibitor Naïve) (N=77) | Total (N=161)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 8 (8)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (6) | 0 (0) | 11 (11) | 15 (18)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Treatment A (Exposed to Ibrutinib) (N=12) | Cohort 1: Treatment B (Exposed to Ibrutinib) (N=41) | Cohort 2: Treatment A (BTK Inhibitor Naïve) (N=31) | Cohort 2: Treatment B (BTK Inhibitor Naïve) (N=77) | Total (N=161)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 8 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 8 (10) | 4 (4) | 6 (9) | 21 (27)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 5 (6) | 11 (12)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 6 (7)
Asthenia (General disorders) | 0 (0) | 7 (7) | 3 (3) | 11 (14) | 21 (24)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4) | 6 (6) | 12 (12)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 2 (3) | 5 (7) | 9 (13)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 6 (6)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (5) | 3 (3) | 12 (13) | 19 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 2 (2) | 12 (13) | 20 (21)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 1 (1) | 7 (7) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 9 (18) | 8 (11) | 26 (40) | 45 (72)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 11 (11)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 6 (6)
Fatigue (General disorders) | 2 (2) | 2 (2) | 2 (2) | 8 (8) | 14 (14)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 8 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 7 (7)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 2 (2) | 3 (6) | 8 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 12 (16) | 13 (17)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 5 (6)
Nasopharyngitis (Infections and infestations) | 2 (3) | 1 (2) | 2 (2) | 3 (4) | 8 (11)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 4 (4) | 8 (8) | 16 (17)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 6 (9) | 3 (4) | 10 (12) | 21 (27)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (9) | 4 (11)
Oedema peripheral (General disorders) | 2 (3) | 3 (4) | 2 (2) | 5 (5) | 12 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 6 (7)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 6 (6) | 9 (10)
Pseudomonas test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 6 (6) | 5 (5) | 12 (15) | 24 (27)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 16 (19) | 23 (26)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 7 (7)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (2) | 0 (0) | 3 (5) | 6 (9)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Testicular oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 2 (2) | 5 (6) | 11 (14)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (4) | 2 (3) | 7 (10)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 9 (9)
Weight decreased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 10 (12) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03235544/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT03235544/SAP_001.pdf